CLINICAL TRIAL: NCT05340829
Title: To Evaluate the Safety, Efficacy, Pharmacokinetics of ThisCART19A in Patients With AIDS Related B Cell Lymphoma/Lympholeukemia
Brief Title: Evaluate the Safety and Effect of ThisCART19A in Patients With AIDS Related B Cell Lymphoma/Lympholeukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: He Huang (Other)
Responsible Party: Sponsor-Investigator, He Huang, President/Proffessor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT400-006
Record Dates: First submitted 2022-04-09; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: AIDS Related Lymphoma and Lympholeukemia
MeSH Terms: conditions — Lymphoma, AIDS-Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ThisCART19A 2×10^6 cells/kg for dose level 1 (Experimental): Patients will receive 2×10^6 cells/kg of ThisCART19A
  Interventions: Biological: ThisCART19A
- ThisCART19A 3×10^6 cells/kg as dose level 2 (Experimental): Patients will receive 3×10^6 cells/kg of ThisCART19A
  Interventions: Biological: ThisCART19A
- Patients will receive 4×10^6 cells/kg as dose level 3 (Experimental): Patients will receive 4×10^6 cells/kg of ThisCART19A
  Interventions: Biological: ThisCART19A

INTERVENTIONS:
Biological: ThisCART19A — ThisCART19A is a new type CAR-T cells therapy for patients with lymphoma and lympholeukemia

SUMMARY:
This is an open label, phase I study to assess the safety and efficacy of ThisCART19A in patients with AIDS related B cell lymphoma/lympholeukemia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Patients with AIDS-associated B-cell lymphoma/leukemia, including but not limited to diffuse large B-cell lymphoma (DLBCL), follicular lymphoma tranferring to DLBCL, mantle cell lymphoma (MCL), follicular lymphoma 3B (FL-3B), original Mediastinal (thymus) large B-cell lymphoma, high-grade B-cell lymphoma and leukemia.
* At least received first line treatment.
* Had available evaluation lesion.
* ECOG(Eastern Cooperative Oncology Group) ≤ 1 or Karnofsky ≥ 60%.
* Had good organic function within 4 weeks before enrollment: Alanine aminotransferase(ALT)≤5×ULN(Upper limit of normal) and total bilirubin(TBIL)<2.0 mg/dL(for patients with Gilbert heald diseases, live involvement and taking atazanavir or indinavir, TBIL<3.0 mg/dL can be enrolled.); Left ventricular ejection fraction(LVEF)≥40%; Absolute neutrophile counts≥1000/mm3; thrombocyte≥30000/mm3; Serum creatinine≤1.5×ULN or creatinine clearance>30 mL/min/1.73 m2.
* Confirmed Cluster of differentiation(CD)19 positive by biopsy for the patients who received CD19 target therapy before.
* Confirmed Human immunodeficiency virus(HIV)-1 infection.
* HIV virus loading < 200 copy/ml within 4 weeks before screening.
* CD4+T cell counts >50 cells/mm3 within 4 weeks before screening.
* Patients with TBIL≤ 1.5 mg/dL, Aspartate aminotransferase(AST) and ALT ≤ 3×ULN, and hepatitis B virus(HBV) DNA <2000 IU/ml can be enrolled for HBV positive patients(defined as hepatitis B virus surface antigen(HBsAg) positive and hepatitis B core(HBc)-total positive ) and hepatitis C virus(HCV) positive patients(defined as HCV antibody positive) . Patients with cirrhosis are excluded.
* Hepatitis B core antibody(HBcAb) positive patients enrolled in this trial have to taking anti-HBV drugs during the whole research.

Exclusion Criteria:

* Known for allergic to the preconditioning measures.
* Uncontrollable bacterial, fungal, viral infection before enrollment.
* Patients with pulmonary embolism within 3 months prior enrollment.
* Intolerable serious cardiovascular and cerebrovascular diseases and hereditary diseases.
* Imaging confirmed the presence of central nervous system involvement(including primary and secondary) and rapid progressing diseases.
* Receive allogeneic hematopoietic stem cell transplantation.
* Systemic steroid use (e.g., prednisone ≥20mg) within 3 days prior to screening. iIntermittent use of topical, inhaled or intranasal steroids recently or currently. Or systemic disease requiring long-term use of immunosuppression drugs.
* Excluded the patients received Influenza vaccinations within 2 weeks prior to lymphodepletion (Received Severe Acute Respiratory Syndrome-Corona virus disease(SARS-COV)19 vaccines could be included. Received inactivated, live/non-live adjuvant vaccines could be enrolled).
* Excluded women who are in pregnant or lactating, and female subjects or partners who plan to be pregnant within 1 year after infusion. Male subjects planning pregnancy within 1 year after infusion should be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity(DLT) observation and the incidence of treatment-emergent adverse events(TEAE) which more than or equal to grade 3 in each dose level | 28 days
  DLT is defined as the incidence of severe adverse events related to ThisCART19A more than 33% in each dose level.

SECONDARY OUTCOMES:
Objective Response rate in patients with AIDS related lymphoma | 12 months
  The incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as best response to treatment
The change characteristics of chimeric antigen receptor(CAR)-T cell number and copy number in patients after infusion | 6 months
  Track CAR-T cells expansion in patients after infusion
Analysis the change characteristics of cytokines and immune effect cells number in patients after infusion | 3 months
  Analysis the effect cells and cytokines in patients after infusion
Analysis the severity and Incidence of Adverse Events in each dose level | 12 months
  Including more than or equal to grade 3 adverse events graded according to the NCI CTCAE v5.0, the adverse events with special consideration
Analysis the immunogenicity(Anti-therapeutic antibody and neutralizing antibody) of CAR-T cells in patients after infusion | 24 months
  Analysis the Anti-therapeutic antibody and neutralizing antibody level after infusion

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, Doctor, Principal Investigator — First hospital affiliated Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China